CLINICAL TRIAL: NCT01094613
Title: MultiCTR Randomized Double-Blind Double-Dummy Study to Evaluate Clinical Efficacy/Safety of DR 6MP for Targeted Ileal Delivery vs Purinethol in Patients w/Moderately Active Crohn's Disease
Brief Title: Multicenter Clinical Efficacy and Safety Study of Delayed Release 6MP in Crohn's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support of study due to reorganization and project prioritization
Sponsor: Teva GTC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol C2/13/DR-6MP-02
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Delayed Release; Targeted Ileal Delivery
MeSH Terms: conditions — Crohn Disease | interventions — Mercaptopurine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Release 6MP (Experimental): 6 Mercaptopurine delayed release oral tablet for targeted ileal delivery, to be administered once nightly before bedtime, for 12 weeks.
  The dose is 2 x 40 mg DR-6MP (total dose, 80 mg DR-6MP).
  Interventions: Drug: Delayed Release 6 mercaptopurine
- Purinethol (Active Comparator): 6 Mercaptopurine Tablet (50 mg) administered orally, at doses of 1-1.5 mg/kg body weight, daily for 12 weeks. Individual patient doses range from 50 mg to 150 mg, including 75, 100 and 125 mg daily, as per patient weight at baseline, and then are up-titrated to clinical efficacy at two week intervals, as needed. Doses may be down-titrated as well if occurrences of AE's warrant dose reduction.
  Interventions: Drug: 6 Mercaptopurine

INTERVENTIONS:
Drug: Delayed Release 6 mercaptopurine — Delayed Release oral tablet for ileal drug delivery, 80 mg, once nightly before bedtime, for 12 weeks.
  Since the study drug must be blinded, patients randomized to this arm will receive the following: 80 mg DR-6MP: 2 active 40 mg DR-6MP tablets.
  Other Names: Delayed Release 6 MP tablet (80 mg)
  Arms: Delayed Release 6MP
Drug: 6 Mercaptopurine — Oral tablet(s) to be administered once daily in the AM, for 12 weeks.Purinethol is available only as a 50 mg tablet; patients randomized to this arm will receive varying doses (dependent on baseline body weight and AE profile) throughout the study;and study drug to be blinded. Therefore, patients randomized to this arm to receive combination active Purinethol/comparable placebo. For ex: 50 mg Purinethol= 1 active 50 mg tablet, 2 comparable placebo tablets; 100 mg Purinethol = 2 active 50 mg tablets, 1 placebo tablet; 150 mg Purinethol = 3 active 50 mg tablets. Patients receiving 75 mg or 125 mg will receive alternating daily doses of 50 and 100 mg, or 100 and 150 mg, respectively, to arrive at a weekly average dose of 75 mg or 125 mg.
  Other Names: Purinethol
  Arms: Purinethol

SUMMARY:
The study is designed to evaluate the clinical efficacy and safety of daily treatment for 12 weeks of oral administration of a delayed release, locally delivered 6MP (mercaptopurine) drug (80 mg), as compared to standard Purinethol (at a dose of 1-1.5 mg/kg/body weight), in alleviating the clinical, immunological and mucosal signs and symptoms of moderately active Crohn's Disease

DETAILED DESCRIPTION:
Crohn's Disease (CD) therapy is aimed at reducing inflammation via induction of remission after a flare-up and maintenance of the remission for as long as possible. Therapies commonly used for inducing remission are steroids and anti-TNF-a. Standard 6MP, on the other hand, has a slow onset of action and requires several months of administration before its therapeutic effects become apparent. Therefore, 6MP is typically used as maintenance therapy, rather than for remission. Furthermore, serious AE's associated wtih 6MP include leucopenia, hepatoxicity, pancreatitis and bone marrow suppression, requiring lowering of dose or treatment discontinuation.

The Teva DR-6MP project was designed to evaluate a new oral 6MP formulation that would address these limitations. The slow action of standard 6MP, precluding its use as a treatment for induction of remission, would be offset by a faster-disintegrating, more soluble formulation with an enteric coating for targeted ileal delivery. This new formulation designed to open at the terminal ileum, the most commonly affected area of CD bowel involvement, could deliver higher effective local concentrations of drug to the site most affected by CD, stimulating an effective local immunological response, resulting in a cascade of widespread immunological activity, evoking an induction of remission. The safety of standard 6MP would be improved upon by the fact that negligible levels of the DR-6MP formulation have been observed in the plasma, obviating the toxicities associated with systemic 6MP. Moreover, since the DR-6MP dose is fixed and not subject to patient weight, nor potentially, side-effects, the dose adjustments required for up-titration to optimal dose, or down-titration due to toxicity, could be avoided.

Previous small, pilot proof-of-concept clinical efficacy and pharmacokinetic studies of the DR-6MP formulation demonstrated the potential for induction of remission, mucosal healing, systemic immunological improvement and lower systemic side-effects.

The current study is designed to repeat the earlier studies under larger, more rigorous conditions in a randomized, double-blind fashion at multiple sites to ascertain if the initial encouraging results could be repeated. Moreover, a higher dose of 6MP (80 mg) will be tested to ascertain if presumably higher local concentrations at the disease site can evince a more robust clinical effect.

ELIGIBILITY:
Inclusion Criteria:

1. Male or (non-pregnant) female, 18-75 years (incl) at screen.
2. Diagnosed w/CD, appropriately documented/supported by endoscopy or radiology.
3. W/ moderately active CD, w/ screen CDAI score 220-450 (inclusive)
4. Screen lab tests:

   * HGB >/= 8.5 g/dL,
   * Platelets >/= 100,000/ mm³
   * WBC >/= 3500 mm³
   * Serum albumin > 2.5 g/dL
   * ALT, AST, ALK Phos, GGTP,. total and direct bilirubin < 2xULN
5. Subjects may be on stable (for at least 2 wks prior screen) 5-ASA, chronic antibiotics or low-dose oral steroids (prednisolone-up to 15 mg daily; budesonide-up to 6 mg daily) and remain on the drug at that dose throughout the study
6. Willing and able to provide written ICF.

Exclusion Criteria:

1. W/ ulcerative colitis or w/ diagnosis of indeterminate colitis.
2. W/ previous bowel resection due to CD resulting in clinically significant Short Bowel Syndrome.
3. W/ fistulizing CD w/ clinic or radiologic evidence of abscess.
4. W/ clinically significant GI obstructive symptoms or x-ray evidence of fibrosed bowel.
5. W/ screen stool culture + for enteric pathogens (Salmonella, Shigella, Campylobacter) or Clostridium difficile toxin assay.
6. W/ hx of persistent intestinal obstruction, bowel perforation, uncontrolled GI bleed,abdominal abscess,infection or toxic megacolon.
7. W/ hx of GI tract malignancy or IBD-associated malignant intestinal changes.
8. W/ surgery/major procedure in 4 weeks prior to 1st study dose.
9. Receiving elemental diet or parenteral nutrition.
10. W/ current signs/symptoms of clinically significant/unstable med/surg condition that precludes safe/complete study participation, determined by med history, PE, ECG, lab tests or imaging. Such conditions may include severe, progressive or uncontrolled renal, metabolic, hepatic, hematologic, endocrine, pulmonary, cardiovascular, psychiatric, neurologic, cerebral or autoimmune disease.
11. W/ serious infections, such as hepatitis, pneumonia, pyelonephritis w/in 12 weeks prior to 1st study dose. Less serious infections such as acute UR tract infections or uncomplicated UT infection not considered exclusions - at discretion of PI.
12. W/ currently known malignancy/pre-malignant lesions/hx of malignancy w/in past 5 years, excl basal cell carcinoma.
13. W/ hx of coagulopathy.
14. W/ porphyria as it may interfere w/ assessment of CD abdominal pain.
15. W/ hx of previous thiopurine failure resulting in serious AE (ex: severe pancreatitis, leucopenia, hepatoxicity or bone marrow suppression) so as to preclude addtl tx w/ 6MP at any dose
16. Taking w/in 6 months prior to 1st study dose (+during study) Active vaccinations (live attenuated bacterial/viral pathogens)
17. Taking w/in 6 weeks prior to 1st study dose (+ during study):

    * Anti-TNFα (infliximab, etanercept, adalimumab)
    * Anti-integrin (natalizumab)
    * Anti-neoplastics, incl methotrexate, daunorubicin hydrochloride
18. Taking w/in 4 weeks prior to 1st study dose (+ during study):

    * Immunosuppressants such as AZA, 6-MP (i.e., other than 6MP drug assigned during study), cyclosporine, tacrolimus, mycophenolate mofetil or thalidomide.
    * Antibiotics or oral/IV corticosteroids (other than oral prednisolone allowed during study as rescue therapy as per protocol).
    * Tx w/ drugs known to induce/inhibit endogenous hepatic drug metabolism such as barbiturates, phenothiazines, cimetidine, carbamazepine etc.
    * Anti-coagulant therapy such as: heparin, warfarin, acenocoumarol.
    * Medications that induce blood dyscrasias or w/ potential for immune dysfunction, bone marrow depression and/or symptoms of CD (diarrhea, abdominal pain).
    * Vaccinations involving inactivated forms of pathogens or purified antigenic proteins (Note: passive immunization involving antibody inoculations permitted at any time)
19. Tx w/in 2 wks prior to 1st study dose (+ during study) IV or oral steroids (prednisolone or budesonide) Antibiotics

    Note: 2 impt exceptions (a) Subjects oral steroid or antibiotic dependent with active CD (CDAI 220-450)in spite of these txs, may remain on tx provided on stable (>=2wks at screen)dose and remain at that dose throughout study (b) Subjects who require steroid-rescue during study
20. Taking w/in 7 days prior to 1st study dose (+ during study):

    * Anticholinergic or other drugs known to affect GI motility.
    * Allopurinol
    * Proton pump inhibitors or other drugs affecting gastric acidity
21. W/body weight below 42.5 kg.
22. Pregnant/nursing at screen, or intend to be during study.
23. Women of childbearing potential not practicing acceptable method of birth control [acceptable methods: surgical sterilization, IUD, contraceptive (oral, patch, or long-acting injectable), partner's vasectomy, double-protection method (condom or diaphragm w/ spermicide) or abstinence].
24. W/ current/hx of drug and/or alcohol abuse.
25. Largely or wholly bed-ridden and w/ little capacity for self-care.
26. W/ known allergy or hypersensitivity to 6-MP or any inactive component of study drug (ex: lactose intolerant).
27. Participated in other clinical trial using investigational drugs w/in 12 weeks prior to 1st study dose.
28. W/ planned elective surgery or hospitalization during study (that may interfere w/ study compliance/outcome).
29. W/inability to communicate well w/investigators/staff (i.e., language problem, poor mental development or impaired cerebral function).
30. Unavailable for trial duration, unable to comply w/schedule, likely to be noncompliant, or felt unsuitable by PI for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with clinical response at study end | 12 weeks
  Clinical response is defined as a reduction in CDAI score (Crohn's Disease Activity Index) by 100 points from baseline, or remission (CDAI score <150),even if it is achieved with reduction of CDAI score of less than 100 points from baseline

SECONDARY OUTCOMES:
Time to clinical response | Week 2, 4, 6, 8 or 12
  Although the primary outcome is to assess the proportion of patients with clinical response at Week 12, we are also interested to see how early during treatment (i.e., between weeks 2 and 12), was this clinical response actually achieved for each treatment group, and if it was maintained until the end of the study (week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Principal Investigator — Hadassah Medical Organization
Locations (11):
- Israel (11):
  - Ha'emek Medical Center, Afula
  - Bnai Zion Hospital, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaarei Tzedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Holy Family Hospital, Nazareth
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh, Ẕerifin

REFERENCES:
- See also: Previous pilot studies (proof of concept efficacy and pk studies) conducted on the DR6MP tablet — http://clinicaltrials.gov